CLINICAL TRIAL: NCT03119402
Title: Combining A Rhythmic Intervention With tDCS to Improve Reading Skills in Dyslexic Adults
Brief Title: Effects of the Combination of RRT With tDCS on Dyslexic Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Alice Cancer, Principal Investigator, Catholic University of the Sacred Heart
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RRT+tDCS
Record Dates: First submitted 2017-04-06; First posted 2017-04-18 (Actual); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Developmental Dyslexia
Keywords: Reading; Developmental Dyslexia; Music; Rhythm; transcranial electrical stimulation; transcranial direct current stimulation
MeSH Terms: conditions — Dyslexia | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants are prevented from having knowledge of which experimental condition (active or sham tDCS) they are assigned to.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- RRT + active tDCS (Experimental): Rhythmic Reading Training, administered for 5 hours over 10 days consecutive (30-minute training sessions per day) + simultaneous 20 minutes of active tDCS (1.5 mA, 5x5cm anodal electrode on left parieto-temporal regions and 5x5cm cathodal electrode on right parieto-temporal regions).
  Interventions: Behavioral: Rhythmic Reading Training; Device: Transcranial direct current stimulation
- RRT + sham tDCS (Sham Comparator): Rhythmic Reading Training, administered for 5 hours over 10 days consecutive (30-minute training sessions per day) + simultaneous 20 minutes of sham tDCS (with the same active tDCS setup, current applied for 30 seconds,
  Interventions: Behavioral: Rhythmic Reading Training; Device: Transcranial direct current stimulation

INTERVENTIONS:
Behavioral: Rhythmic Reading Training — RRT is a computerized reading training program designed for Italian students with dyslexia. The main feature of this intervention is the integration of a traditional remediation approach (sublexical treatment) with rhythm processing. Therefore, all reading exercises are characterized by a rhythmic accompaniment with gradually increasing speed.
  Other Names: RRT
Device: Transcranial direct current stimulation — tDCS (transcranial direct current stimulation) is a noninvasive weak-current brain stimulation technique that can facilitate (anodal electrode) or inhibit (cathodal electrode) cortical activity, thus offering exciting possibilities for the enhancement and treatment of impaired cognitive abilities.
  Other Names: tDCS

SUMMARY:
The purpose of the study is to evaluate the effectiveness of the combination of Rhythmic Reading Training (RRT), a computer-assisted intervention method that combines sublexical reading exercises with rhythm processing, and transcranial direct current stimulation (tDCS) on reading abilities of a group of Italian undergraduate students with dyslexia. Two experimental conditions (active vs. sham) will be compared. Finally, the effects of the intervention on other cognitive functions involved in the process of reading (i.e., rapid automatized naming, verbal working memory, rhythm perception abilities) will be measured.

ELIGIBILITY:
Inclusion Criteria:

* having been diagnosed with DD (ICD-10 code: F81.0) on the basis of standard inclusion and exclusion criteria (ICD-10: World Health Organization, 1992) and of the diagnosis procedure followed in the Italian practice

Exclusion Criteria:

* presence of comorbidity with other neuropsychiatric or psychopathological conditions (whereas comorbidity with other learning disabilities were allowed)
* exclusion criteria for the use of tDCS (e.g. epilepsy, pregnancy).

Ages: 19 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-04-18 (Actual); Primary Completion 2017-09-04 (Actual); Study Completion 2018-04-04 (Estimated)

PRIMARY OUTCOMES:
Text reading speed expressed in syllables per seconds | 2 weeks
  The ability to read aloud a text was assessed using the Italian standardized test 'Prova di velocità di lettura di brani' (Zoccolotti, Fondazione S. Lucia), which provides speed and accuracy scores in reading aloud age-normed texts.
Text reading accuracy expressed in number of errors | 2 weeks
  The ability to read aloud a text was assessed using the Italian standardized test 'Prova di velocità di lettura di brani' (Zoccolotti, Fondazione S. Lucia), which provides speed and accuracy scores in reading aloud age-normed texts.
Word reading speed expressed in syllables per seconds | 2 weeks
  The ability to read aloud lists of words was assessed using the following Italian standardized tests: 'Assessment battery for Developmental Dyslexia and Dysorthography-2' (Batteria per la valutazione della dislessia e disortografia evolutiva - DDE-2), in which speed and accuracy scores were computed for word reading (4 lists of 28 words each with different lengths and frequency of use); 'Word and pseudo-word reading test' (WPRT, Prova di lettura di parole e non parole), in which speed and accuracy scores were computed for word reading (4 lists of 30 words varying according to length: short vs. long and frequency of use: low vs. high frequency).
Word reading accuracy expressed in number of errors | 2 weeks
  The ability to read aloud lists of words was assessed using the following Italian standardized tests: 'Assessment battery for Developmental Dyslexia and Dysorthography-2' (Batteria per la valutazione della dislessia e disortografia evolutiva - DDE-2), in which speed and accuracy scores were computed for word reading (4 lists of 28 words each with different lengths and frequency of use); 'Word and pseudo-word reading test' (WPRT, Prova di lettura di parole e non parole), in which speed and accuracy scores were computed for word reading (4 lists of 30 words varying according to length: short vs. long and frequency of use: low vs. high frequency).
Pseudo-word reading speed expressed in syllables per seconds | 2 weeks
  The ability to read aloud lists of pseudo-words was assessed using the following Italian standardized tests: 'Assessment battery for Developmental Dyslexia and Dysorthography-2' (Batteria per la valutazione della dislessia e disortografia evolutiva - DDE-2), in which speed and accuracy scores were computed for pseudo-word reading (2 lists of 16 pseudo-words each with different lengths); 'Word and pseudo-word reading test' (WPRT, Prova di lettura di parole e non parole), in which speed and accuracy scores were computed for pseudo-words reading (2 lists of 30 pseudo-words varying for length: short vs. long).
Pseudo-word reading accuracy expressed in number of errors | 2 weeks
  The ability to read aloud lists of pseudo-words was assessed using the following Italian standardized tests: 'Assessment battery for Developmental Dyslexia and Dysorthography-2' (Batteria per la valutazione della dislessia e disortografia evolutiva - DDE-2), in which speed and accuracy scores were computed for pseudo-word reading (2 lists of 16 pseudo-words each with different lengths); 'Word and pseudo-word reading test' (WPRT, Prova di lettura di parole e non parole), in which speed and accuracy scores were computed for pseudo-words reading (2 lists of 30 pseudo-words varying for length: short vs. long).

SECONDARY OUTCOMES:
Rapid Automatized Naming | 2 weeks
  Rapid Automatized Naming of colours and figures
Verbal Working Memory | 2 weeks
  Onwards and backwards digit span
Rhythm Discrimination | 2 weeks
  Rhythm discrimination task

CONTACTS AND LOCATIONS:
Locations (1):
- Catholic University of the Sacred Heart, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided